CLINICAL TRIAL: NCT00065260
Title: A Randomized Trial of Immunosuppression in Aplastic Anemia Patients With Refractory Pancytopenia or Suboptimal Hematologic Response After h-ATG/CsA Treatment
Brief Title: Rabbit Antithymocyte Globulin Versus Campath-1H for Treating Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030249; 03-H-0249
Record Dates: First submitted 2003-07-18; First posted 2003-07-21 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Aplastic Anemia
Keywords: Alemtuzumab (Campath-1H); Rabbit ATG; Severe Aplastic Anemia; Cyclosporine; Thrombocytopenia; Leukopenia; Neutropenia; Autoimmunity; Relapse; Anemia
MeSH Terms: conditions — Anemia, Aplastic; Thrombocytopenia; Leukopenia; Neutropenia; Autoimmune Diseases; Recurrence; Anemia | interventions — Alemtuzumab; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- r-ATG /cyclosporine (Experimental): A randomized trial of rabbit anti-thymocyte globulin (r-ATG)/ cyclosporine (CsA) versus Campath-1H in aplastic anemia patients with refractory pancytopenia or suboptimal hematological response after horse ATG treatment. Subjects who receive rabbit ATG/ CsA will be given rabbit ATG 3.5mg/kg/day for 5 days and CsA 10mg/kg/day orally twice daily for 6 months (15mg/kg/day for children under 12 yrs. Subjects who receive Campath-1H will receive an intravenous infusion for 10 days. Adult subjects will receive 10mg/day (children:0.2mg/kg/day).
  Interventions: Drug: r-ATG; Drug: CsA
- Alemtuzumab (Campath-1H) (Experimental): A randomized trial of rabbit anti-thymocyte globulin (ATG)/ cyclosporine (CsA) versus Campath-1H in aplastic anemia patients with refractory pancytopenia or suboptimal hematological response after horse ATG treatment. Subjects who receive rabbit ATG/ CsA will be given rabbit ATG 3.5mg/kg/day for 5 days and CsA 10mg/kg/day orally twice daily for 6 months (15mg/kg/day for children under 12 yrs. Subjects who receive Campath-1H will receive an intravenous infusion for 10 days. Adult subjects will receive 10mg/day (children:0.2mg/kg/day).
  Interventions: Drug: Campath-1H

INTERVENTIONS:
Drug: Campath-1H — Campath-1H IV 10 days. Adults:10mg/day (children:0.2mg/kg/day).
  Other Names: Alemtuzumab
  Arms: Alemtuzumab (Campath-1H)
Drug: r-ATG — Rabbit ATG 3.5mg/kg/day for consecutive 5 days
  Other Names: Rabbit Anti-Thymoglobulin
  Arms: r-ATG /cyclosporine
Drug: CsA — CsA 10mg/kg/day orally twice daily for 6 months (15mg/kg/day for children under 12 yrs.
  Other Names: Cyclosporine
  Arms: r-ATG /cyclosporine

SUMMARY:
Severe aplastic anemia, characterized by pancytopenia and a hypocellular bone marrow, is effectively treated by immunosuppressive therapy, usually a combination of antithymocyte globulin (ATG) and cyclosporine (CsA). Survival rates following this regimen are equivalent to those achieved with allogeneic stem cells transplantation. However, approximately 1/3 of patients will not show blood count improvement after ATG/CsA. General experience and small pilot studies have suggested that such patients may benefit from further immunosuppression. Furthermore, analysis of our own clinical data suggest that patients with poor blood count responses to a single course of ATG, even when transfusion-independence is achieved, have a markedly worse prognosis than patients with robust hematologic improvement. The management of such cases is uncertain.

This study will enroll patients who are either refractory to h-ATG (continued severe pancytopenia) or who have only modest improvement in blood counts (weak hematologic responders) to receive a further immunosuppressive therapy, delivered either as rabbit ATG (Thymoglobulin, r-ATG) or a humanized monoclonal antibody to T-cells, alemtuzumab (Campath-1H ). Primary endpoint will be response rate at 3 months defined as no longer meeting criteria for severe aplastic anemia. Relapse, robustness of hematopoietic recovery at 3 months, survival and clonal evolution to paroxysmal nocturnal hemoglobinuria (PNH), myelodysplasia and acute leukemia will be the secondary endpoints.

DETAILED DESCRIPTION:
Severe aplastic anemia, characterized by pancytopenia and a hypocellular bone marrow, is effectively treated by immunosuppressive therapy, usually a combination of antithymocyte globulin (ATG) and cyclosporine (CsA). Survival rates following this regimen are equivalent to those achieved with allogeneic stem cells transplantation. However, approximately 1/3 of patients will not show blood count improvement after ATG/CsA. General experience and small pilot studies have suggested that such patients may benefit from further immunosuppression. Furthermore, analysis of our own clinical data suggest that patients with poor blood count responses to a single course of ATG, even when transfusion-independence is achieved, have a markedly worse prognosis than patients with robust hematologic improvement. The management of such cases is uncertain.

This study will enroll patients who are either refractory to h-ATG (continued severe pancytopenia) or who have only modest improvement in blood counts (weak hematologic responders) to receive further immunosuppressive therapy, delivered either as rabbit ATG (Thymoglobulin , r-ATG) or a humanized monoclonal antibody to T-cells, alemtuzumab (Campath-1H ). Primary endpoint will be response rate at 6 months defined as no longer meeting criteria for severe aplastic anemia. Relapse, robustness of hematopoietic recovery at 6 months, survival and clonal evolution to paroxysmal nocturnal hemoglobinuria (PNH), myelodysplasia and acute leukemia will be the secondary endpoints.

ELIGIBILITY:
* INCLUSION CRITERIA:

Severe aplastic anemia confirmed at NIH by:

Bone marrow cellularity less than 30% (excluding lymphocytes)

At least two of the following:

Absolute neutrophil count less than 500/microL;

Platelet count less than 20,000/ microL;

Reticulocyte count less than 60,000/ microL.

Severe aplastic anemia refractory to prior course(s) of h-ATG/CsA defined after 3 months from treatment with less or equal to 4 years from receiving h-ATG.

OR

Suboptimal response to initial immunosuppression with h-ATG/CsA as defined by platelet and reticulocyte count less than 50,000 /microL at 3 months.

Age greater than or equal to 2 years of age

EXCLUSION CRITERIA:

Diagnosis of Fanconi anemia.

Evidence of a clonal disorder on cytogenetics. Patients with super severe neutropenia (ANC less than 200/microL) will not be excluded initially if results of cytogenetics are not available or pending. If evidence of a clonal disorder is later identified, the subject will go off study.

Prior treatment courses with rabbit ATG or high dose cyclophosphamide (200 mg/kg or equivalent).

Infection not adequately responding to appropriate therapy.

Underlying immunodeficiency state including seropositivity for HIV.

Failure to discontinue the herbal supplements Echinacea purpurea or Usnea barbata (Old Man's Beard) within two weeks of enrollment.

Previous hypersensitivity to Campath-1H or its components.

Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy or that death within 7-10 days is likely.

Potential subjects with cancer who are on active chemotherapeutic treatment or who take drugs with hematological effects will not be eligible.

Serum creatinine greater than 2.5 mg/dL.

Current pregnancy or lactation or unwillingness to take contraceptives.

Inability to understand the investigational nature of the study or give informed consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-11-06 (Actual); Primary Completion 2010-12-29 (Actual); Study Completion 2016-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Townsley, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS, Maciejewski J. The pathophysiology of acquired aplastic anemia. N Engl J Med. 1997 May 8;336(19):1365-72. doi: 10.1056/NEJM199705083361906. No abstract available. PMID 9134878
- [Background] Mathe G, Amiel JL, Schwarzenberg L, Choay J, Trolard P, Schneider M, Hayat M, Schlumberger JR, Jasmin C. Bone marrow graft in man after conditioning by antilymphocytic serum. Br Med J. 1970 Apr 18;2(5702):131-6. doi: 10.1136/bmj.2.5702.131. PMID 4909449
- [Background] Stein RS, Means RT Jr, Krantz SB, Flexner JM, Greer JP. Treatment of aplastic anemia with an investigational antilymphocyte serum prepared in rabbits. Am J Med Sci. 1994 Dec;308(6):338-43. doi: 10.1097/00000441-199412000-00005. PMID 7985721
- [Derived] Scheinberg P, Nunez O, Weinstein B, Scheinberg P, Wu CO, Young NS. Activity of alemtuzumab monotherapy in treatment-naive, relapsed, and refractory severe acquired aplastic anemia. Blood. 2012 Jan 12;119(2):345-54. doi: 10.1182/blood-2011-05-352328. Epub 2011 Nov 8. PMID 22067384
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-H-0249.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | r-ATG /Cyclosporine | Alemtuzumab (Campath-1H)
Started | 27 | 27
Completed | 27 | 26
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | r-ATG /Cyclosporine | Alemtuzumab (Campath-1H) | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 9 | 12
  Between 18 and 65 years | 22 | 14 | 36
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Participants no Longer Meeting Criteria for Severe Aplastic Anemia.
Description: Number of participants no longer meeting the criteria for severe aplastic anemia as measured by response to treatment at 6 months
Time Frame: 6 months
Population: 1 patient was not evaluable at 6 months in the alemtuzumab arm because of a single early death from infectious complications
Measure: Number; unit: participants
Arm/Group | r-ATG /Cyclosporine | Alemtuzumab (Campath-1H)
Number analyzed (Participants) | 27 | 26
participants
  No Response | 18 | 17
  Partial Response | 9 | 9
  Complete Response | 0 | 0

2. Secondary Outcome: Number of Participants With Robust Hematologic Recovery With Reticulocyte or Platelet Count
Description: Number of participants with robust hematologic recovery with reticulocyte or platelet count ≥ 50,000/uL
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | r-ATG /Cyclosporine | Alemtuzumab (Campath-1H)
Number analyzed (Participants) | 27 | 26
Participants | 9 | 9

3. Secondary Outcome: Percentage of Cumulative Incidence of Relapse in Participants
Description: Percentage of cumulative incidence of relapse of disease in participants
Time Frame: 3 year
Population: 1 participants was not evaluable at 6 months in the alemtuzumab arm because of a single early death from infectious complications.
Measure: Number; unit: percentage of cumulative incidence
Arm/Group | r-ATG /Cyclosporine | Alemtuzumab (Campath-1H)
Number analyzed (Participants) | 27 | 26
percentage of cumulative incidence | 19 | 9

4. Secondary Outcome: Percentage of Cumulative Incidence of Clonal Evolution in Participants
Description: Percent of cumulative incidence of clonal evolution in participants to either paroxysmal nocturnal hemoglobinuria (PNH), myelodysplasia or acute leukemia.
Time Frame: 3 years
Population: 1 participant was not evaluable at 6 months in the alemtuzumab arm because of a single early death from infectious complications
Measure: Number; unit: Percentage of Cumulative Incidence
Arm/Group | r-ATG /Cyclosporine | Alemtuzumab (Campath-1H)
Number analyzed (Participants) | 27 | 26
Percentage of Cumulative Incidence | 16 | 5

5. Secondary Outcome: Percentage of Participants no Longer Meeting Criteria for Severe Aplastic Anemia.
Description: Percentage of participants no longer meeting the criteria for severe aplastic anemia as measured by response to treatment
Time Frame: 3 months and 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | r-ATG /Cyclosporine | Alemtuzumab (Campath-1H)
Number analyzed (Participants) | 27 | 26
percentage of participants
  3 Months | 19 [3 to 34] | 19 [3 to 34]
  6 Months | 33 [14 to 52] | 37 [18 to 57]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | r-ATG /Cyclosporine | Alemtuzumab (Campath-1H)
All-Cause Mortality (participants affected / at risk) | 9/27 | 4/27
Serious Adverse Events (participants affected / at risk) | 7/27 | 12/27
Other Adverse Events (participants affected / at risk) | 7/27 | 12/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | r-ATG /Cyclosporine (N=27) | Alemtuzumab (Campath-1H) (N=27)
infection (Immune system disorders) | 7 (7) | 12 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | r-ATG /Cyclosporine (N=27) | Alemtuzumab (Campath-1H) (N=27)
infection (Blood and lymphatic system disorders) | 7 (7) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes